CLINICAL TRIAL: NCT05369754
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of YBSW015 Injection in Healthy Subjects
Brief Title: A Phase Ia Clinical Study to Evaluate the Safety, Tolerability, PK and Immunogenicity of YBSW015 in Healthy Subjects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yabao Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: YBSW015001
Record Dates: First submitted 2022-04-30; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YBSW015 injection 180mg (Experimental)
  Interventions: Biological: YBSW015 injection
- YBSW015 injection 450mg (Experimental)
  Interventions: Biological: YBSW015 injection
- YBSW015 injection 900mg (Experimental)
  Interventions: Biological: YBSW015 injection
- YBSW015 injection 1800mg (Experimental)
  Interventions: Biological: YBSW015 injection

INTERVENTIONS:
Biological: YBSW015 injection — Prepared YBSW015 injection is intravenously injected by an infusion pump or gravity infusion with intravenous infusion of 250 mL for 60 min±10 min.

SUMMARY:
This is phase Ia study to research YBSW015 injection which is a monomolecular bispecific antibody. The Primary objective is to evaluate the safety and tolerability of YBSW015 injection after a single intravenous injection at different doses in healthy subjects.

The Secondary objective is to evaluate the pharmacokinetic characteristics and immunogenicity of different doses of YBSW015 injection after a single intravenous injection in healthy subjects. This study is a single-center, randomized, double-blind, placebo-controlled, single-dose escalation clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and ≤ 55 years at screening, regardless of gender;
2. Body weight ≥50kg for males and ≥45kg for females, body mass index (BMI) between 18.0 kg/m2and 30.0 kg/m2 (inclusive) at screening;
3. Subject who has negative result in the YBSW015 serology test in screening;
4. Has completed COVID-19 vaccination and the last dose more than 6 weeks prior to randomization
5. Subject who are normal in the physical examination, vital signs, laboratory tests and other auxiliary examinations (chest radiograph, abdominal ultrasound scan, 12-lead ECG, etc.), or abnormal without clinical significance as judged by the investigator;
6. Subject who has a negative result in the urine human chorionic gonadotropin test in screening period, and a negative result in the blood human chorionic gonadotropin test in baseline period;
7. Subjects (including their partners) who do not have a pregnancy plan and are willing to adopt effective contraception measures from signing the informed consent to 6 months after administration of the investigational drug;
8. Subjects who has understood the trial feature, significance, possible benefits, possible inconveniences and potential risks and discomforts in detail, and are willing to participate in this clinical trial and are able to communicate well with the investigator and follow the requirements of the entire study, and has signed the written informed consent form prior to the trial.

Exclusion Criteria:

1. The positive results are obtained in SARS-CoV-2 nucleic acid test using nasal swabs prior to screening and randomization (results within 7 days prior to randomization);
2. Has recent SARS-CoV-2 infection that resolved within 6 weeks prior to randomization；
3. Those who have received any SARS-CoV-2 immunoglobulin, plasma from COVID-19 survivors in recovery period（within 15 weeks）;
4. Those who have used therapeutic biologics within 12 weeks before screening, or those who are in drug elimination period currently (within 5 half-lives), whichever is longer;
5. Those who have participated in clinical study of other intervention investigational products within 12 weeks prior to screening, or those who are in drug elimination period currently (within 5 half-lives), whichever is longer;
6. Those who have been vaccinated against pathogens other than SARS CoV-2 within 6 weeks prior to screening, or plan to be vaccinated against pathogens other than SARS CoV-2 during the study or within 6 weeks after the study;
7. Those who have taken herbal medicines, dietary supplements (excluding vitamin, mineral and trace element supplements), or any prescription or non-prescription drugs within 14 days (inclusive) prior to screening;
8. Those who have had major surgery history within 8 weeks (including 8 weeks) before screening, or plan to perform surgeries during the study, and those who are exposed to unacceptable risks brought by such surgery at the discretion of the sponsor and the investigator;
9. Those who have an abnormal electrocardiogram with clinical significance at screening, or QTc> 450 msec, or other abnormal electrocardiogram data with clinical significance;
10. Subjects with poor blood pressure control (systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg);
11. Positive serology test results for hepatitis C virus antibody, human immunodeficiency virus antibody, Syphilis Treponema Pallidum antibody (S-TP) and hepatitis B virus surface antigen (HBsAg) at Screening;
12. Those who have a history of transplantation in vital organs (such as heart, lung, liver and kidney);
13. Patients with malignant tumors (excluding those whose malignant tumors have been cured with no recurrence in recent 5 years, with complete excision of skin basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of any type);
14. Those who have cardiovascular diseases, respiratory diseases, gastrointestinal diseases, endocrine system diseases, hematological system diseases or nervous system diseases, and are exposed to higher risks by taking the investigational drug, or those whose disease state can obviously change absorption, distribution, metabolism or excretion of the investigational drug;
15. Those who have a history of drug abuse or drug taking within 5 years prior to screening or have a positive result in urine drug test;
16. Those who have a history of alcoholism or excessive drinking (14 units of alcohol per week :1 unit = 285 mL beer, or 25 mL liquor, or 100 mL wine) within 6 months prior to screening or have a positive result in alcohol breath test;
17. Those who smoke ≥5 cigarettes per day within 6 months prior to screening, or are unwilling/unable to stop nicotine intake during the study;
18. Those who are known to be allergic to the investigational drug, monoclonal antibody drug, therapeutic protein preparation, human serum albumin, cytokines, interleukin etc. or have a history of or a propensity to allergy;
19. Females with a positive result of pregnancy test and lactating females;
20. Those who have a blood loss or donation of greater than 400 mL, or received blood transfusion or blood products within the past 3 months, or plan to donate blood during the study;
21. Those with a history of needle sickness, hemophobia or intolerance of venipunctures;
22. Subjects who cannot complete the study due to other reasons or are supposed to be excluded at the discretion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
safety of YBSW015 injection | from screening visit to the end of the follow-up period, assessed up to 85 days
  Evaluation of treatment-emergent adverse event (TEAE) and serious adverse events (SAE) during treatment;
tolerability of YBSW015 injection | from screening visit to the end of the follow-up period, assessed up to 85 days
  Evaluation of local tolerance: administration site reaction;

SECONDARY OUTCOMES:
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  Peak concentration (Cmax) Immunogenicity: To detect the positive rate and titer of anti-drug antibody ADA
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  peak time (Tmax)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  terminal elimination rate constant (λz)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  terminal elimination half-life (t1/2)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  area under the curve from time zero to the time of the last time of quantifiable concentration (AUC0-t)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  area under the concentration-time curve from time zero to infinite time (AUC0-∞)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  extrapolated percentage of AUC0-∞ (%AUCex)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  apparent clearance (CLz)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  apparent volume of distribution (Vz)
PK parameter | from screening visit to the end of follow-up period, assessed up to 85 days
  mean residence time (MRT)
Immunogenicity | from screening visit to the end of follow-up period, assessed up to 85 days
  positive rate of anti-drug antibody ADA
Immunogenicity | from screening visit to the end of follow-up period, assessed up to 85 days
  Titer of anti-drug antibody ADA

IPD SHARING:
Plan to Share IPD: No